CLINICAL TRIAL: NCT00535197
Title: A Phase I/II Safety and Tolerability Study Following the Autologous Infusion of Immuno-selected CD34+ Subset Bone Marrow Stem Cells Into Patients With Acute Total Anterior Circulation Ischaemic Stroke
Brief Title: Autologous Bone Marrow Stem Cells in Ischemic Stroke.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HHSC/003
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Stroke, Acute; Infarction, Middle Cerebral Artery
Keywords: Stroke; Middle Cerebral Artery
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD34+ stem/progenitor cell therapy (Experimental): Patients presenting within 7 days of onset with severe anterior circulation ischemic stroke (National Institutes of Health Stroke Scale [NIHSS] score≥8). CD34+ cells were collected from the bone marrow of the subjects before being delivered by catheter angiography into the ipsilesional middle cerebral artery.
  Interventions: Biological: Infusion of autologous CD34+ stem cells into middle cerebral artery

INTERVENTIONS:
Biological: Infusion of autologous CD34+ stem cells into middle cerebral artery — intra-arterial infusion into ipsilateral MCA, via trans-femoral approach

SUMMARY:
The aim of the study is to determine the safety and tolerability of an autologous CD34+ subset bone marrow stem cell infusion into the middle cerebral artery in patients who have suffered acute total or partial anterior circulation syndrome (TACS/PACS).

DETAILED DESCRIPTION:
The proposed trial will involve the recruitment of a total of 10 patients.

The cells will be collected from each subject recruited, via bone marrow sampling. CD34+ stem cells will then be isolated and harvested during a process of immuno-selection in accordance with the principles of Good Manufacturing Practice. The CD34+ cells will then be directly infused into the area of the stroke intra-arterially using the middle cerebral artery.

Initially, the investigator will monitor each patient for a period of 6 months post-stem cell infusion. Thereafter, they will revert to their previous treatment regime in the clinic.

Assessment of adverse events will be by physical examination and measurement of laboratory parameters. Assessment of efficacy will be by physical examination and the measurement of laboratory, CT and MRI parameters.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of clinically definite acute stroke
* Time of stroke onset is known and treatment can be started within 7 days of onset
* CT or MRI brain scanning has reliably excluded both intracranial haemorrhage and structural brain lesions which can mimic stroke (e.g. cerebral tumour)
* The stroke is severe and conforming to the TACS phenotype (weakness, homonymous hemianopia and a focal cognitive deficit (e.g. aphasia) or reduction in consciousness) or PACS phenotype (two out of the three TACS criteria)
* An age range of 30-80 years old
* Stroke confined to MCA territory on CT or MRI brain imaging
* NIHSS score >/= 8

Exclusion Criteria:

* Known defect of clotting or platelet function (but patients on anti-platelet agents can enrol)
* Haematological causes of stroke
* Severe co-morbidity
* Hepatic or renal dysfunction
* The patient is female and of childbearing potential (unless it is certain that pregnancy is not possible) or breast feeding
* Hypo- or hyperglycaemia sufficient to account for the neurological symptoms; the patient should be excluded if their blood glucose is < 3.0 or > 20.0mmol/L
* Patient is likely to be unavailable for follow-up e.g. no fixed home address
* Patients with evidence of life threatening infection (e.g. HIV) or life threatening illness (e.g. advanced cancer)
* Patient was already dependent in activities of daily living before the present acute stroke
* Patients who have been included in any other clinical trial within the previous month

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety will be evaluated in terms of adverse events graded according to CTC toxicity criteria and laboratory test results | Duration of study
  safety will be evaluated in terms of adverse events graded according to CTC toxicity criteria and laboratory test results

SECONDARY OUTCOMES:
Improvement in clinical function as assessed by the Modified Rankin Score, and NIH stroke scale. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Habib, Professor, Principal Investigator — Imperial College London U.K.
Locations (1):
- St Marys Hospital, Paddington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banerjee S, Bentley P, Hamady M, Marley S, Davis J, Shlebak A, Nicholls J, Williamson DA, Jensen SL, Gordon M, Habib N, Chataway J. Intra-Arterial Immunoselected CD34+ Stem Cells for Acute Ischemic Stroke. Stem Cells Transl Med. 2014 Nov;3(11):1322-30. doi: 10.5966/sctm.2013-0178. Epub 2014 Aug 8. PMID 25107583
- [Derived] Mackie AR, Losordo DW. CD34-positive stem cells: in the treatment of heart and vascular disease in human beings. Tex Heart Inst J. 2011;38(5):474-85. PMID 22163120